CLINICAL TRIAL: NCT00501696
Title: A Randomized Placebo-Controlled, Crossover-Design Study of the Effects of Low Dose Naltrexone on Quality of Life as Measured by the Multiple Sclerosis Quality of Life Inventory (MSQLI54)
Brief Title: A Randomized Placebo-Controlled, Crossover-Design Study of the Effects of Low Dose Naltrexone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: UCSF MS Center, UCSF MS Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H43034-30200-02
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2007-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Naltrexone; Cross-Over Studies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): A randomized placebo-controlled, parallel-group study, crossover-design
  Interventions: Drug: 4.5 mg Naltrexone; Drug: Naltrexone
- 2 (Other): A randomized placebo-controlled, parallel-group study, crossover-design
  Interventions: Drug: 4.5 mg Naltrexone

INTERVENTIONS:
Drug: 4.5 mg Naltrexone — low dose naltrexone 4,5mg on the multiple sclerosis quality of life inventory (MSQLI54)
  Other Names: Naltrexon(4.5mg) or placebo , crossover-design
Drug: Naltrexone — 4,5mg low dose naltrexone on the multiple sclerosis quality of life inventory (MSQLI54)
  Other Names: Naltrexone(4.5mg) or placebo , crossover-design
  Arms: 1

SUMMARY:
This is a randomized placebo-controlled, parallel-group study, crossover-design of the effects of low dose naltrexone on the multiple sclerosis quality of life inventory (MSQLI54)

This study will assess the impact of LDN compared to placebo on quality of life as measured by the composite score of the MSQOL54 in adult subjects with MS.

Also we plan:

1. To compare the 10 scales of the MSQOL54 during the active treatment and placebo cycles between active treatment and placebo groups
2. To compare each individual's composite response to LDN versus placebo during the active treatment and placebo cycles
3. To compare each individual on the 10 scales of the MSQOL54 during the active treatment and placebo cycles

DETAILED DESCRIPTION:
Immunomodulatory and immunosuppressive therapies are known to modify the course of the disease. Interferon beta-1a, interferon beta-1b and glatiramer acetate are immunomodulators whereas mitoxantrone and natalizumab are immunosuppressants

The disease modifying therapies decrease the frequency of relapses and are associated with improved neurological outcomes relative to placebo. However, these medications are only partially effective, are expensive, require either frequent self injections or intravenous infusion and have significant side effects. None are proven in the progressive forms of MS and none of alleviate the symptoms associated with MS.

Endogenous Opioid peptides and Naltrexone:

Low dose naltrexone (LDN) is proposed to adjust the level of endorphins in the body thereby enhancing immune function and is anecdotally beneficial in MS. LDN is inexpensive, easily administered (one capsule a day at bedtime), and virtually has no serious side effect (during the first weeks of LDN use, some patients complain of some difficulty sleeping, that rarely persists after the first week). Although use of LDN is popular within the MS community efficacy is not proven because clinical trials have not been performed.

Naltrexone, is an opioid antagonist approved by the FDA in 1984 in a 50mg dose for the treatment of opioid and alcohol abuse. By blocking opioid receptors, naltrexone also blocks reception of the endogenous opioid peptides: beta-endorphin, metenkephalin and dynorphin. Virtually every cell of the immune system has receptor for these mediators. These peptides regulate a wide range of biological activities, including immune responses through interaction with G-protein coupled transmembrane opioid receptors.

In 1985, Bernard Bihari, MD, described the effects of low dose Naltrexone (1.5-4.5 mg Naltrexone) on the body's immune system. He discovered that people with HIV had less than twenty percent of the normal level of endorphins. He began looking for ways to raise endorphin without blocking its receptors and found that 1.75-4.5 mg Naltrexone (Low Dose Naltrexone, LDN) at bed time raises the endorphin level up to 100 to 300 percent during the night. Dr. Bihari has reported beneficial effects of LDN on a variety of diseases such as cancers (e.g. Multiple Myeloma, Lymphoma, Hodgkin's disease, breast cancer, GI cancers, non small cell cancer of lung, malignant melanoma, neuroblastoma, ovarian cancer, prostate cancer, renal cell carcinoma, and uterine cancer), amyotrophic lateral sclerosis, Alzheimer's disease, Behçet's disease, celiac disease, chronic fatigue syndrome, Crohn's disease, emphysema, fibromyalgia, HIV/AIDS, Irritable bowel syndrome, Parkinson's disease, pemphigoid, psoriasis, multiple sclerosis, rheumatoid arthritis, systemic Lupus erythematosus, ulcerative colitis and Wegner's granulomatosis . Despite these anecdotal claims there are no published studies demonstrating efficacy of LDN in any disease state.

Because of its low cost and ease of administration and anecdotal reports of efficacy LDN has gained a significant gross-roots following among patients and doctors. There are some striking reports about beneficial effects of LDN on relapse reduction and disability and in general patients treated with LDN report improvements in a sense of well being, fatigue, as well as bowel, bladder and sexual function.

Immunological Mechanisms Involved in MS and effects of LDN β-endorphin is an opioid peptide, synthesized by cells of the central nervous system (arcuate nucleus) and immune system (lymphocytes, thymocytes, monocytes and splenocytes). This peptide is decreased in concentration in peripheral blood mononuclear cells (PBMC) of MS patients, with the lowest concentrations linked to the progressive forms of the disease. Furthermore increased concentrations of β-endorphin are found during interferon beta treatment and following clinical relapses. In the animal model of MS, experimental autoimmune encephalitis, β-endorphin blockade worsens disability.

Lesions in MS may be the result of oligodendroglial apoptosis and microglial activation rather than neuroinflammatory processes. Activated microglia secrete proinflammatory and neurotoxic factors (nitric oxide and peroxynitrites) that could cause neurodegeneration. In theory, inhibition of microglia would be protective in MS. Naltrexone, is capable of reducing microglial cytokine (IL-1β) and nitric oxide in glial cultures. If naltrexone is beneficial in MS, a possible mechanism of action is through reduction in microglial nitric oxide synthase activity resulting in decreased peroxynitrites production. Peroxynitrites are thought to inhibit glutamate transporters thereby increasing the synaptic concentrations of glutamate resulting in excitatory neurotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS by current International Criteria
* Between 18 and 75 years of age
* Willingness to not change or start disease modifying or symptomatic therapies of MS during the trial
* The patient should be able to understand English
* The patients should read, understand and sign the study informed consent form prior to any participation in the study
* Patients currently on a disease modifying therapy should be on this medication for at least 3 months and not anticipate changing or discontinuing this medication during the 17 week study
* Patients not currently on a disease modifying therapy
* For women of childbearing potential, willingness to use a barrier method of contraception during the trial

Exclusion Criteria:

* Start of a disease modifying therapy within 3 months of entry in the trial
* Planned start of DMT during the clinical trial
* Pregnancy
* Current chronic opioid agonists use, i.e. any narcotic medication including hydroxycode and codeine-containing preparations
* Patients under 18 years of age
* Patients older than 75 years prior to the start of therapy
* Patients who are currently on both interferon and glatiramer acetate
* Patients who are currently taking LDN
* Patients who are currently taking immunosuppressive medications e.g. cyclophosphamide, mitoxantrone, azathioprine, methotrexate, mycophenolate mofetil, natalizumab, rituximab, alemtuzumab or other immune suppressants
* Participation in other clinical treatment trials in MS
* The patients who cannot comprehend MSQLI54 instructions and

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
comparison of the mean score between treated and placebo groups, adjusting for differences in the baseline score between the two groups; comparison of each of the 10 scales of the MSQLI54 between treated and placebo groups | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kornyeyva, MD, PhD, Principal Investigator — MS Center , UCSF
Locations (1):
- MS Center UCSF, Parnassus Ave, suite #908, San Francisco, California, United States